CLINICAL TRIAL: NCT00245128
Title: A Phase II Pilot Study to Determine the Safety and Preliminary Efficacy of Imatinib Mesylate (Gleevec) in Patients With Myelofibrosis With Myeloid Metaplasia
Brief Title: Imatinib Mesylate in Treating Patients With Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per PI, results from another similar study were published prior to study analysis. Negative study results were published therefore analysis was not completed
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445435; OHSU-541 (Other: OHSU IRB); OHSU-HEM-01071-L (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Myeloproliferative Disorders
Keywords: chronic idiopathic myelofibrosis; polycythemia vera; essential thrombocythemia
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: imatinib mesylate — Once daily oral administration of Imatinib Mesylate at a dose of 600mg for 12 months.

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying the side effects of imatinib mesylate and how well it works in treating patients with myelofibrosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety, efficacy, and tolerability of imatinib mesylate in patients with myelofibrosis with myeloid metaplasia.
* Determine the 3-, 6-, and 12-month major and minor erythroid response rates in patients treated with this drug.

Secondary

* Determine reduction in marrow fibrosis in patients treated with this drug.
* Determine decrease in spleen size in patients treated with this drug.

OUTLINE: This is a multicenter, open-label, nonrandomized, pilot study.

Patients receive oral imatinib mesylate once daily for 1 year in the absence of disease progression or unacceptable toxicity. Patients who do not experience a minor erythroid response or a 50% reduction in spleen size after 6 months of treatment are removed from the study. Patients experiencing clinical benefit (e.g., ongoing erythroid response) after 1 year of treatment may continue treatment with imatinib mesylate as above at the discretion of the principal investigator.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelofibrosis with myeloid metaplasia (MMM), defined by all of the following:

  * Leukoerythroblastic blood picture
  * Fibrosis involving > 1/3 sectional area of bone marrow biopsy
  * Splenomegaly (unless patient has undergone prior splenectomy)
  * Philadelphia chromosome negative
  * No myelodysplastic syndrome
  * No systemic disorders associated with marrow fibrosis
* Red blood cell transfusion dependent, defined by 1 of the following:

  * Patient has required ≥ 2 units of red blood cells every 4 weeks within the past 8 weeks
  * Hemoglobin ≤ 8 g/dL on ≥ 3 occasions (≥ 2 weeks apart ) over the past 8 weeks
* No evidence of disease transformation to acute myelogenous leukemia, defined as > 20% blasts in bone marrow and/or peripheral blood

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 50,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 2 times ULN (unless due to extramedullary hematopoiesis in the liver)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No New York Heart Association grade III-IV heart disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier method contraception during and for 3 months after completion of study treatment
* No serious, uncontrolled medical condition
* No patients who are considered potentially unreliable or with a history of noncompliance to medical regimens

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 2 weeks since prior interferon alfa

Chemotherapy

* No concurrent chemotherapy except hydroxyurea to control elevated blood counts

Endocrine therapy

* More than 4 weeks since prior corticosteroids, danazol, or other androgens for MMM

Other

* More than 4 weeks since other prior treatment for MMM
* No other concurrent experimental drug therapy for MMM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2007-03 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mauro, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib Mesylate (Gleevec): Once daily oral administration of Imatinib Mesylate at a dose of 600mg for 12 months.
Period: Overall Study
Arm/Group | Imatinib Mesylate (Gleevec)
Started | 10
Completed | 0
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate (Gleevec)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 68.2 (11.00303)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major and/or Minor Erythroid Responses at 3, 6, and 12 Months of Therapy
Description: A major response = transfusion independent or a>2.0g/dl rise in hemoglobin without transfusion maintained for at least 8 weeks.
  Minor response= > 1 to 2.0g/dl incremental rise in hemoglobin maintained for at lease 8 weeks with a decrease in transfusion requirements of at least 50% compared to the mean transfusion requirement during the 8 week pre-study period.
Time Frame: At 3,6, and 12 months of therapy
Measure: Number; unit: percentage of participants
Arm/Group | Imatinib Mesylate (Gleevec)
Number analyzed (Participants) | 0

2. Secondary Outcome: Reduction in Marrow Fibrosis and Decrease in Spleen Size
Time Frame: After 6 and 12 months of therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Imatinib Mesylate (Gleevec)
Serious Adverse Events (participants affected / at risk) | 10/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate (Gleevec) (N=10)
Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 2
Hypersensitivity Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Spontaneous Abortion (Reproductive system and breast disorders) | 2
Elevated CPK (Blood and lymphatic system disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Parkinson's Disease (Nervous system disorders) | 1
Liver abscess (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute leukemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Oesophageal adenocarcinoma (Respiratory, thoracic and mediastinal disorders) | 1
Optic nerve atrophy (Eye disorders) | 1
hospitalization for bone pain (Musculoskeletal and connective tissue disorders) | 1
Oncocytoma (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Extra pyramidal symptoms (Nervous system disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Lower abdominal pain (Gastrointestinal disorders) | 1
Ureteric Calculus (Renal and urinary disorders) | 1
Bacterial meningitis (Infections and infestations) | 1
Bilirubin and lipase (Renal and urinary disorders) | 1
ateriovenus malformation (Vascular disorders) | 1
Cholelithiasis (Renal and urinary disorders) | 1
Esophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Hypocalcemia (Blood and lymphatic system disorders) | 1
Hodgkin's Disease (Blood and lymphatic system disorders) | 1
Retinal detachment (Eye disorders) | 1
Fatal diverticulitis, gastrointestinal peforation, peritonitis (Gastrointestinal disorders) | 1
Fatal pancreatitis (Gastrointestinal disorders) | 1
Prostate Cancer (Reproductive system and breast disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Ptosis (Eye disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1
Death (General disorders) | 1 — Disease progression
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Brain herniation (Nervous system disorders) | 1
Priapism (Reproductive system and breast disorders) | 1
Squamous cell carcinoma of the penis (Reproductive system and breast disorders) | 1
Leydig cell hyperplasia (Reproductive system and breast disorders) | 1
Urothelial Carcinoma (Renal and urinary disorders) | 1
Bell's Palsy (Nervous system disorders) | 1
Plaques of demyelination (Nervous system disorders) | 1
Interstitial nephritis (Renal and urinary disorders) | 1
Hemorrhagic cystitis (Renal and urinary disorders) | 1
Metastases of breast cancer (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (Gleevec) (N=10)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination/results were never analyzed due to negative study results from other similar studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No